CLINICAL TRIAL: NCT03783052
Title: Gastrointestinal Physiological Conditions in Obesity and After Bariatric Surgery
Acronym: GASTON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S60930
Record Dates: First submitted 2018-08-10; First posted 2018-12-20 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Healthy volunteers (Other): 11 Healthy volunteers
  Interventions: Device: SmartPill in fasted state; Device: SmartPill in fed state
- Obese volunteers (Other): 11 Obese Volunteers
  Interventions: Device: SmartPill in fasted state; Device: SmartPill in fed state
- Roux-en-Y Gastric Bypass patients (Other): 6 volunteers with a Roux-en-Y Gastric Bypass
  Interventions: Device: SmartPill in fasted state; Other: Aspiration; Other: Gastric emptying scintigraphy
- Sleeve Gastrectomy patients (Other): 6 volunteers with a Sleeve Gastrectomy
  Interventions: Device: SmartPill in fasted state; Other: Aspiration; Other: Gastric emptying scintigraphy
- Volunteers with obesity (Other): 6 obese volunteers
  Interventions: Device: SmartPill in fasted state; Other: Aspiration; Other: Gastric emptying scintigraphy

INTERVENTIONS:
Device: SmartPill in fasted state — SmartPill administration in fasted state
Device: SmartPill in fed state — SmartPill administration in fed state
  Arms: Healthy volunteers; Obese volunteers
Other: Aspiration — Aspiration of gastrointestinal samples in fasted and fed state
  Arms: Roux-en-Y Gastric Bypass patients; Sleeve Gastrectomy patients; Volunteers with obesity
Other: Gastric emptying scintigraphy — Gastric emptying scintigraphy in fed state
  Arms: Roux-en-Y Gastric Bypass patients; Sleeve Gastrectomy patients; Volunteers with obesity

SUMMARY:
Over the years, obesity has become a major public health concern. The increasing rates of obesity are associated with an enhanced demand for weight-loss with bariatric surgery as a treatment option. Bariatric surgery procedures alter the anatomical structure of the gastrointestinal tract, which contributes to the postoperative weight loss. However, it is not sure how obesity and the anatomical alterations of bariatric surgery affect the gastrointestinal physiology including gastrointestinal pH, gastric emptying, intestinal transit time and concentration of enzymes.

DETAILED DESCRIPTION:
During the visit in the obesity clinic, eligible patients will be approached for participation by the sub-investigator. Interested patients will receive information regarding the study and receive the information sheet containing the informed consent form. After signing the informed consent form, volunteers will be invited to come to the clinical research center:

* Healthy volunteers: Gastrointestinal physiology will be analyzed during two visits using a telemetric capsule. During the first visit, the physiological conditions of interest will be analysed in fasted state using the telemetric capsule. During the second visit, the physiological conditions of interest will be analysed in fed state using the telemetric capsule.
* Obese volunteers: Gastrointestinal physiology will be analyzed during two visits using a telemetric capsule. During the first visit, the physiological conditions of interest will be analysed in fasted state using the telemetric capsule. During the second visit, the physiological conditions of interest will be analysed in fed state using the telemetric capsule.
* Obese volunteers: Gastrointestinal physiology will be analyzed during three visits using a telemetric capsule, scintigraphy and via the collection of gastrointestinal samples. During the first visit, the physiological conditions of interest will be analysed in fasted state using the telemetric capsule. During the second visit, gastrointestinal samples will be collected at the level of the stomach, the duodenum and jejunum via aspiration through multiple lumen catheters in fasted and fed state. During the third visit, gastric emptying will be observed via scintigraphy in fed state.
* Volunteers after Sleeve Gastrectomy: Gastrointestinal physiology will be analyzed during three visits using a telemetric capsule, scintigraphy and via the collection of gastrointestinal samples. During the first visit, the physiological conditions of interest will be analysed in fasted state using the telemetric capsule. During the second visit, gastrointestinal samples will be collected at the level of the sleeve, the duodenum and jejunum via aspiration through multiple lumen catheters in fasted and fed state. During the third visit, gastric emptying will be observed via scintigraphy in fed state.
* Volunteers after Roux-en-Y gastric Bypass: Gastrointestinal physiology will be analyzed during three visits using a telemetric capsule, scintigraphy and via the collection of gastrointestinal samples. During the first visit, the physiological conditions of interest will be analysed in fasted state using the telemetric capsule. During the second visit, gastrointestinal samples will be collected at the level of the pouch, the Roux limb and the common limb via aspiration through multiple lumen catheters in fasted and fed state. During the third visit, gastric emptying will be observed via scintigraphy in fed state.

ELIGIBILITY:
Inclusion Criteria:

- 18 years or older

Exclusion Criteria:

* History of gastric ulcers
* Disorders of swallowing
* Suspected strictures, fistulas or physiological GI obstruction.
* GI surgery within past three months
* Severe dysphagia to food or pills
* Crohns disease or diverticulitis
* Use of implanted or portable electro-mechanical medical devices
* Known intolerance to the SmartPill device
* Known food allergies to any component of the meal
* History of multiple bariatric surgeries
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Temperature | 0-7 days
  Gastrointestinal Temperature (°C)
Gastrointestinal pH | 0-7 days
  Gastrointestinal pH (pH values)
Gastrointestinal Pressure | 0-7 days
  Gastrointestinal Pressure (mmHg)
Concentration of bile acids | 1 day
  Concentration of bile acids
Gastric emptying time | 2 hours
  Gastric emptying time

SECONDARY OUTCOMES:
Gastrointestinal motility | 0-7 days
  Contractions per minute
Gastrointestinal transit times | 0-7 days
  Gastric Emptying Time (hours), Small Bowel Transit Time (hours), Colonic Transit Time (hours) and Whole Gut Transit Time (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Van der Schueren, PhD, Principal Investigator — UZ Leuven, Department of Endocrinology
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No